CLINICAL TRIAL: NCT04299620
Title: Micro-Ultrasound to Whole Mount Image Correlation for Detection and Localization of Prostate Cancer
Brief Title: Micro-Ultrasound for the Detection and Localization of Prostate Cancer Tumors in Patients Undergoing Radical Prostatectomy
Status: Active, not recruiting | Phase: Not Applicable | Type: Interventional
Sponsor: Jonsson Comprehensive Cancer Center (Other)
Collaborators: Exact Imaging (Industry); Phase One Foundation (Other)
Responsible Party: Sponsor
Allocation: Not Applicable | Model: Single Group | Masking: None | Purpose: Diagnostic
Other Study IDs: 19-001136; NCI-2019-05784 (Registry Identifier: CTRP (Clinical Trial Reporting Program)); 19-001136 (Other: UCLA / Jonsson Comprehensive Cancer Center)
Record Dates: First submitted 2020-02-19; First posted 2020-03-09 (Actual); Last update posted 2023-10-06 (Actual); Status verified 2022-10

CONDITIONS: Prostate Carcinoma
MeSH Terms: conditions — Prostatic Neoplasms | interventions — Ultrasound, High-Intensity Focused, Transrectal

STUDY DESIGN:
Oversight: Data Monitoring Committee: Yes | FDA-regulated Drug: No | FDA-regulated Device: Yes | US Export: No

ARMS (1):
- Diagnostic (TRUS) (Experimental): Patients may undergo TRUS prior to standard-of-care radical prostatectomy. Following radical prostatectomy, removed glands are scanned and micro-US, standard of care mpMRI, and whole mount images are analyzed and compared.
  Interventions: Device: Digital Image Analysis; Procedure: Radical Prostatectomy; Procedure: Transrectal Ultrasound

INTERVENTIONS:
Device: Digital Image Analysis — Analysis of images
Procedure: Radical Prostatectomy — Undergo standard of care radical prostatectomy
  Other Names: Prostatovesiculectomy
Procedure: Transrectal Ultrasound — Undergo transrectal ultrasound
  Other Names: endorectal ultrasound; ERUS (endorectal ultrasound); TRUS

SUMMARY:
This trial studies the ability of micro-ultrasound to detect and characterize prostate cancer tumors in patients undergoing radical prostatectomy (removal of the entire prostate and some of the tissue around it). Usually multiparametric magnetic resonance imaging is used for the detection and targeted therapy of prostate cancer, but its accuracy remains imperfect. Micro-ultrasound may be superior as it provides real-time tumor visualization which may simplify and improve prostate cancer targeted therapy. This may also reduce the need for and substantial costs of radical prostatectomy.

DETAILED DESCRIPTION:
PRIMARY OBJECTIVE:

I. Determine if micro-ultrasound (US) can be used to identify prostate cancer foci with equivalent (non-inferior) performance relative to multiparametric magnetic resonance imaging (mpMRI).

SECONDARY OBJECTIVE:

I. Determine if micro-US can be used to contour prostate cancer foci with equivalent (non-inferior) accuracy to mpMRI.

TERTIARY OBJECTIVE:

I. Determine if ex vivo micro-US images have quality comparable to in vivo micro-US images.

QUATERNARY OBJECTIVE:

I. Determine if micro-US can be used to evaluate suspicion of extracapsular extension (ECE) with equivalent (non-inferior) accuracy to mpMRI.

OUTLINE:

Patients may undergo transrectal micro-ultrasound scan (TRUS) prior to standard-of-care radical prostatectomy. Following radical prostatectomy, removed glands are scanned and micro-US, standard of care mpMRI, and whole mount images are analyzed and compared.

ELIGIBILITY:
Inclusion Criteria:

* Standard-of-care mpMRI within the past 12 months
* Biopsy-proven prostate cancer, Gleason grade >= 3+3
* Maximum posterior-to-anterior prostate dimension of =< 6 cm
* Scheduled to receive standard-of-care radical prostatectomy

Exclusion Criteria:

* Maximum posterior-to-anterior prostate dimension greater than 6 cm
* Prior radiation or focal treatment for prostate cancer
* Inability to have a transrectal ultrasound scan
* Prostate biopsy < 4 weeks prior to surgery

Min Age: 18 Years | Sex: Male | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 86 (Actual)
Dates: Start 2020-10-21 (Actual); Primary Completion 2022-06-14 (Actual); Study Completion 2025-09-01 (Estimated)

PRIMARY OUTCOMES:
Identification of prostate cancer foci | Up to 3 years
  Will be evaluated by comparing sensitivity and positive predictive value of multiparametric magnetic resonance imaging (mpMRI) and micro-ultrasound (US) for identification of prostate cancer (CaP) foci.
  Measurement tool = chi squared test

SECONDARY OUTCOMES:
Contours of prostate cancer foci | Up to 3 years
  evaluated by measuring the dice similarity coefficient (DSC) and Hausdorff distances (Hd) between micro-ultrasound (US) and whole mount (WM) tumor contours, and between mpMRI and WM tumor contours. The difference between tumor diameter and volume will be computed between WM and mpMRI, and between WM and US. All measures will then be used to compare accuracy of US versus mpMRI.
  Wilcoxon signed-rank tests:
  Signed rank tests are nonparametric matched pair tests, here mostly used to compare correlation of mpMRI and WM v. correlation of US and WM. Minimum and maximum input values will depend on the metric being tested; min and max output values will vary between zero and one. A higher output indicates less difference in performance between mpMRI and US. A lower score indicates that more a difference between mpMRI and US. Whether a lower score is a better outcome or worse outcome depends on which modality (mpMRI vs US) is more strongly correlated with WM.

OTHER OUTCOMES:
Ex vivo and in vivo micro-US images | Up to 3 years
  Differences in in vivo versus ex vivo image quality will be evaluated by testing for systematic differences in tumor contouring accuracy. The measures will be identical to those listed under "secondary outcome measures" above, but for comparison between ex vivo micro ultrasound and in vivo micro ultrasound (instead of MRI).
Suspicion of extracapsular extension (ECE) | Up to 3 years
  Micro ultrasound and mpMRI ECE suspicion scores will be compared for ECE-positive tumors. Micro ultrasound and mpMRI ECE suspicion scores will also be compared for ECE-negative tumors.
  Measurement tool(s) = Wilcoxon signed-rank test and one-sided non-inferiority t-test.
  Notes on the use of Wilcoxon signed-rank tests: (see outcome 2 description above)

CONTACTS AND LOCATIONS:
Overall Officials: Leonard S Marks, Principal Investigator — UCLA / Jonsson Comprehensive Cancer Center
Locations (1):
- UCLA / Jonsson Comprehensive Cancer Center, Los Angeles, California, United States